CLINICAL TRIAL: NCT00581256
Title: A Randomized Comparison of Radiation Therapy Techniques in the Management of Node Positive Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2004.038; IRB #2002-387 ~ HUM 39607 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Results first posted 2016-12-01 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
Keywords: left sided
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Best Delivery-optimized radiotherapy technique (IMRT)
  Interventions: Radiation: IMRT
- 2 (Active Comparator): Best 3-dimensional standard PWTF technique
  Interventions: Radiation: 3D

INTERVENTIONS:
Radiation: IMRT — All patients treated with the optimized plan will be treated to the entire target volume to 52.2 Gy in 1.74 Gy fractions, which is biologically equivalent to 50 Gy in 2 Gy fractions. This fractionation scheme will allow the boost of 10 Gy to be incorporated into the planning directive and to be delivered simultaneously with the treatment to the remaining target volume.
  Arms: 1
Radiation: 3D — All patients treated using the best standard technique will receive 50 Gy in 2 Gy fractions or 50.4 Gy in 1.8 Gy fractions to the entire target volume delivering one treatment per day, five fractions per week (excluding holidays). A boost of 10 Gy to the tumor bed of an intact breast will be delivered. Patients treated to the chest wall will receive a 10Gy scar boost if mastectomy margins are positive in a patient with Stage II disease or if the patient was originally diagnosed with T3 or T4 (Stage III) disease
  Arms: 2

SUMMARY:
Radiotherapy has been shown to reduce breast-cancer specific mortality in patients at high risk for distant dissemination. It has also been shown to increase rates of non-breast cancer deaths and morbidity due to cardiovascular and pulmonary toxicity. Although treatment planning has improved significantly through the years, recent reports still demonstrate treatment-related morbidity even with 3-dimensional planned techniques. Thus, while 3D planning represents the state of the art treatment for loco-regional radiotherapy for breast cancer, further improvement is needed to continue to decrease heart and lung exposure. The ultimate goal of the proposed research is to determine whether treatment planning using intensity-modulated radiotherapy (IMRT), the "next generation" of radiation treatment delivery systems, results in less radiation exposure to the heart and lungs than the best current RT technique in women with node positive breast cancer. This proposal will test the potential clinical value of IMRT compared to the best standard 3D plan (partially wide tangent fields, PWTF) in the treatment of breast cancer. These two treatment techniques will be studied in a Phase II randomized trial using quantitative indicators of potential cardiac and lung toxicity. The preliminary data generated from this trial will be used to ultimately justify a multi-institutional comparison of the two treatment techniques with long-term clinical cardiac and pulmonary toxicity as endpoints.

DETAILED DESCRIPTION:
1. Primary Objective 1.1 To compare the extent of new myocardial perfusion defects following breast cancer radiotherapy using the best standard 3-D radiotherapy technique, partially wide tangent fields, versus the best optimized technique.
2. Secondary Objectives 2.1 To compare changes in ejection fraction and alterations in cardiac wall motion with treatment by technique 2.2 To compare changes in lung perfusion defects and pulmonary function tests (DLCO, FEV1, and FVC) by technique 2.3 To compare rates of pericarditis and pneumonitis by technique

Cardiac Endpoints: Myocardial SPECT-CT perfusion defects, ejection fraction, alterations in cardiac wall motion, per SPECT-CT (adenosine stress and rest (if necessary)) scan.

Pulmonary Endpoints: Lung SPECT-CT perfusion defects per SPECT-CT scan, and changes in pulmonary function tests: DLCO, FEV1, FVC Clinical Endpoints: pericarditis and pneumonitis.

ELIGIBILITY:
Inclusion Criteria:

Eligibility Criteria

* Breast cancer diagnosis: Patients must have histologically confirmed adenocarcinoma of the breast requiring comprehensive loco-regional irradiation that includes treatment to the intact breast/chest wall, supraclavicular (SCV), infraclavicular nodes (ICV), and internal mammary nodes (IMN).
* Patients must have pathologic T 1, 2, 3 or 4, N 1, 2, or 3 Stage II or III disease as defined by the AJCC Staging System, 6th edition. Patients who do not undergo axillary staging but are at risk for nodal involvement may also be treated.
* All patients must have left-sided breast cancer.
* Both men and women are eligible.
* Patients must be adults (18 years of age or older)
* For women of child-bearing age, effective contraception must be used. A written statement must be obtained that the patient is not pregnant. If there is any question of pregnancy at time of therapeutic RT or at time of each SPECT-CT scan, a pregnancy test will be done to confirm the patient is not pregnant.
* Performance status should be 0-2 by ECOG criteria.
* Patients that have received prior RT may be enrolled on the present study if the new breast lesion can be treated with no overlap of RT fields.
* Patients must be aware of the neoplastic nature of her/his disease.
* Patients must be informed of the investigational nature of this study and must sign an informed consent in accordance with the Institutional Review Board (IRB) of the University of Michigan and federal guidelines.
* Patients' blood tests should indicate they are able to tolerate radiotherapy. Tests must be done within 28 days of registration:

CBC with differential and platelet count (Hemoglobin > 8.0 g/dl; wbc > 2000/mm3; absolute neutrophil count > 1000/mm3; platelet count > 75,000/mm3.

Exclusion Criteria:

* Patients who are pregnant or are nursing are excluded.
* Pathologically node negative breast cancer unless treated with neo-adjuvant chemotherapy.
* Performance status > 2 by ECOG criteria
* Patients who are unable to lie on their back and raise their arm above their head in the treatment planning position for radiotherapy
* Patients with a clinically unstable medical condition
* Patients with a life-threatening disease state
* History or suspicion of serious life-threatening allergic reaction to Tc-99m imaging agents.
* Patients that have had breast-conservation surgery with positive margins or any patient with negative margins with a tumor positive for an extensive intraductal component.
* Patients that are not able to use the ABC device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-04; Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Pierce, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Jagsi R, Griffith KA, Moran JM, Ficaro E, Marsh R, Dess RT, Chung E, Liss AL, Hayman JA, Mayo CS, Flaherty K, Corbett J, Pierce L. A Randomized Comparison of Radiation Therapy Techniques in the Management of Node-Positive Breast Cancer: Primary Outcomes Analysis. Int J Radiat Oncol Biol Phys. 2018 Aug 1;101(5):1149-1158. doi: 10.1016/j.ijrobp.2018.04.075. Epub 2018 May 5. PMID 30012527

RESULTS

PARTICIPANT FLOW:
Groups:
- IMRT: Best Delivery-optimized radiotherapy technique (IMRT)
  IMRT: All patients treated with the optimized plan will be treated to the entire target volume to 52.2 Gy in 1.74 Gy fractions, which is biologically equivalent to 50 Gy in 2 Gy fractions. This fractionation scheme will allow the boost of 10 Gy to be incorporated into the planning directive and to be delivered simultaneously with the treatment to the remaining target volume.
- 3DRT: Best 3-dimensional standard PWTF technique
  3D: All patients treated using the best standard technique will receive 50 Gy in 2 Gy fractions or 50.4 Gy in 1.8 Gy fractions to the entire target volume delivering one treatment per day, five fractions per week (excluding holidays). A boost of 10 Gy to the tumor bed of an intact breast will be delivered. Patients treated to the chest wall will receive a 10Gy scar boost if mastectomy margins are positive in a patient with Stage II disease or if the patient was originally diagnosed with T3 or T4 (Stage III) disease
Period: Overall Study
Arm/Group | IMRT | 3DRT
Started | 28 | 26
Completed | 28 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IMRT | 3DRT | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Continuous [Mean (Full Range); unit: years] | 47.8 [30 to 69] | 51.7 [25 to 74] | 50.6 [25 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With a Significant Increase in Perfusion Defects (PD)
Description: To compare the extent of new myocardial perfusion defects following breast cancer radiotherapy using the best standard 3-D radiotherapy technique, partially wide tangent fields, versus the best optimized technique. Perfusion defects (PD) were assessed by comparing normalized perfusion distributions against our institution's normal polar map databases for the left anterior descending artery (LAD) using thresholds of 2.5-SD (standard deviation) and 1.5-SD below the normal mean. On the basis of interest variability, a PD increase greater than 5% or 10% was considered significant for 2.5- and 1.5-SD thresholds, respectively.
Time Frame: 1 Year
Measure: Number; unit: participants
Arm/Group | IMRT | 3DRT
Number analyzed (Participants) | 28 | 26
participants
  2.5 SD and PD increase >5% | 1 | 2
  1.5 SD and PD increase >10% | 3 | 5
Statistical Analysis 1: Comparison: IMRT vs 3DRT; A Perfusion Defect (PD) increase of greater than 5% for a 2.5 SD threshold was considered significant; Test type: Superiority or Other; p = 0.6, Fisher Exact
Statistical Analysis 2: Comparison: IMRT vs 3DRT; A PD increase of greater than 10% for a 1.5 SD threshold was considered significant; Test type: Superiority or Other; p = 0.46, Fisher Exact

2. Secondary Outcome: Mean Percent Change in Ejection Fraction (LVEF)
Description: To compare change in ejection fraction between treatment arms.
Time Frame: baseline to approx 1 year
Measure: Mean (Full Range); unit: percent change
Arm/Group | IMRT | 3DRT
Number analyzed (Participants) | 28 | 26
percent change | 3 [-7 to 18] | -2 [-16 to 11]

3. Secondary Outcome: Number of Participants With New Lung Perfusion Defects
Description: To compare changes in lung perfusion defects by treatment arm. Perfusion defects (PD) were assessed by comparing normalized perfusion distributions against our institution's normal polar map databases for the left anterior descending artery (LAD).
Time Frame: baseline to approx 1 year
Population: One patient randomized to the IMRT arm did not receive her post-RT lung SPECT scan therefore pre- and post-radiotherapy Lung SPECT scans were available for 53 patients.
Measure: Number; unit: participants
Arm/Group | IMRT | 3DRT
Number analyzed (Participants) | 27 | 26
participants | 3 | 5

4. Secondary Outcome: The Number of Participants That Experience Pericarditis and Pneumonitis
Description: To compare rates of pericarditis and pneumonitis by treatment arm.
  Pericarditis (inflammation of the pericardium):
  Grade1: Asymptomatic, ECG or physical exam; changes consistent with pericarditis Grade 2: Symptomatic pericarditis Grade 3: Pericarditis with physiologic consequences Grade 4: Life-threatening Pneumonitis (inflammation of the walls of the alveoli in the lungs) Grade 1: Asymptomatic, radiographic findings only Grade 2: Symptomatic, not interfering with ADL (activities of daily living) Grade 3: Symptomatic, interfering with ADL Grade 4: Life-threatening
Time Frame: approx 1 year
Measure: Number; unit: participants
Arm/Group | IMRT | 3DRT
Number analyzed (Participants) | 28 | 26
participants
  Number of participants with pericarditis (Gr 1-4) | 0 | 0
  Number of participants with pneumonitis (Gr 1-4) | 0 | 0

ADVERSE EVENTS:
Arm/Group | IMRT | 3DRT
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/26
Other Adverse Events (participants affected / at risk) | 27/28 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT (N=28) | 3DRT (N=26)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 | 0 — ANC (Absolute Neutrophil Count), grades range from 1-5 where 1 is mild elevation and 5 is death)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT (N=28) | 3DRT (N=26)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Breast nipple/areolar deformity (Reproductive system and breast disorders) | 4 | 5
Breast volume/hypoplasia (Reproductive system and breast disorders) | 9 | 7
Burn (Skin and subcutaneous tissue disorders) | 1 | 4
Cardiac General - Other (Cardiac disorders) | 0 | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 3
Edema: limb (Vascular disorders) | 10 | 11
Edema: trunk/genital (Vascular disorders) | 1 | 2
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 0 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9 | 12
Fibrosis-deep connective tissue (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 0 | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flashes/flushes (General disorders) | 1 | 2
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 22 | 17
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 11 | 8
Infection with Grade 3 or 4 neutrophils (Infections and infestations) | 0 | 1
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 0 | 1
Joint-function (Musculoskeletal and connective tissue disorders) | 0 | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 1
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 | 1
Lymphatics - Other (Blood and lymphatic system disorders) | 0 | 1
Lymphedema-related fibrosis (Blood and lymphatic system disorders) | 2 | 4
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1
Mood alteration (Psychiatric disorders) | 2 | 2
Muscle weakness, generalized (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Neuropathy: motor (Nervous system disorders) | 1 | 1
Pain (General disorders) | 7 | 7
Pain - Other (General disorders) | 1 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 4
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 | 2
Rash: dermatitis associated with radiation (Skin and subcutaneous tissue disorders) | 11 | 16
Seroma (Injury, poisoning and procedural complications) | 1 | 1
Sexual/Reproductive Function - Other (Reproductive system and breast disorders) | 1 | 1
Sodium, serum-low (hyponatremia) (Investigations) | 1 | 1
Telangiectasia (Vascular disorders) | 9 | 4
Tremor (Nervous system disorders) | 1 | 1
Vaginal dryness (Reproductive system and breast disorders) | 1 | 1
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 2 | 0
Atrophy, skin (Skin and subcutaneous tissue disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Creatinine (Investigations) | 1 | 0
Dermal change lymphedema, phlebolymphedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 2 | 0
Neuropathy: sensory (Nervous system disorders) | 1 | 1
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes